CLINICAL TRIAL: NCT02638363
Title: An Investigation of General Predictors for Cognitive Behavioral Therapy Outcome for Anxiety Disorders in a Naturalistic Setting
Brief Title: An Investigation of General Predictors for CBT Outcome for Anxiety Disorders in a Naturalistic Setting
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Sara Kerstine Kaya Nielsen, PhD Student, Clinical Psychologist, University of Copenhagen
Other Study IDs: Precat
Record Dates: First submitted 2015-12-16; First posted 2015-12-23 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — The participants will receive 12-16 sessions of manualized group-based CBT with a maximum of 8 participants in each group. The therapists are trained psychiatrists, psychologists, or nurses under supervision. The treatment manuals are developed by mental health professionals in the Capital Region of Denmark. The treatment program includes traditional CBT components (e.g., psychoeducation, identification of thoughts and feelings, exposure, cognitive restructuring, and relapse prevention).

SUMMARY:
The aim of this study is to investigate the predictive value of emotion regulation and attentional control for outcome of Cognitive Behavioural Therapy for adults with anxiety disorders in a naturalistic setting.

DETAILED DESCRIPTION:
Anxiety disorders are a pervasive problem, with an estimated 12-month prevalence of 16.6 %, and they are associated with significant impairment and high social costs. Cognitive behavioral therapy (CBT) has shown to be effective and for treating of anxiety disorders. CBT is furthermore cost-effectiveness.This has made CBT the first choice of treatment for anxiety disorders in many mental health settings around the world. Despite this impressive evidence-base, a relatively large group of individuals do not benefit from CBT, relapse, or drop out of treatment. Thus, there is a clear and pressing need to improve the efficacy and effectiveness of CBT for anxiety disorders. One way in which to improve is to identify predictors of CBT outcome. In naturalistic clinical settings, identification of prognostic factors can help allocate resources to those presumed to benefit most from CBT, while also identifying those who may need additional CBT, adjunctive therapy, or entirely different treatment to maximize outcomes.

Current knowledge about who is most likely to benefit from CBT is sparse and stems primarily from well-controlled laboratory settings. These results may not generalize to patient outcomes in mental health settings, in which patients with more severe and comorbid disorders are often seen. Thus, naturalistic studies have the potential to significantly increase knowledge, inform clinical strategies, and thus improve the treatment offered in mental health settings. Furthermore, existing studies have mostly investigated socio-demographic factors as predictors of drop-out and non-response. However, these variables have shown to be either non-significant or inconsistent predictors of outcome. Results concerning comorbidity as a predictor are also mixed. In sum, knowledge on who is most likely to benefit from CBT is sparse, and to date no reliable predictors have been identified.

While prior work has primarily emphasized atheoretical predictors, it may prove more fruitful to focus on predictor variables stemming from psychological theories. Identifying such predictors can provide direct prognostic information for clinicians. Additionally, these predictors could also inform the development of adjunctive components of treatment that may optimize the treatment for those with poorer CBT outcome. Some exciting studies suggest that such a line of inquiry could yield relevant results.

Maintaining factors is one aspect highlighted by several therapeutic approaches/theories as crucial for the treatment of anxiety disorders, and accordingly these factors are often the target of cognitive and behavioral treatments. Emotion regulation and attentional control are examples of key maintaining factors in anxiety disorders. CBT, which aims to teach patients cognitive reappraisal of maladaptive cognitions and encourages approach (rather than avoidance) behavior via cognitive restructuring and exposure, may be more suitable for patients with certain characteristics. Specifically, recent research and theory suggest that it is crucial for effective treatment of anxiety disorders that clients learn to tolerate fear while being exposed to anxiety-provoking stimuli, rather than merely habituating to the stimuli. Learning to tolerate fear may require emotion regulation skills and the ability to control attention and this has been supported by recent studies. However, so far only certain areas of emotion regulation have been investigated and to date never in a naturalistic setting. Attentional control has never been examined as a predictor of CBT outcomes. Accordingly, this study is designed to investigate the predictive value of attentional control and of three facets of emotion regulation skills.

Attentional control There is strong evidence that individuals with anxiety disorders have biased attention towards threatening stimuli, but there is no consensus as to why these biases occur. Recent research suggests that it is not the threat bias per se that is problematic. Rather, individual differences in the ability to voluntarily control attention may affect the impact of threatening information hence increasing or decreasing the anxiety symptoms. A potential consequence may be that individuals with low ability to voluntarily control their attention have difficulties participating in exposure and/or do not progress in the exposure hierarchy, because the level of anxiety gets too high. This may subsequently lead to failure to learn that fear is not dangerous or even drop-out of CBT. Furthermore, a pronounced bias towards irrelevant negative information may take up so many resources that processing of important, relevant information is hampered, making it difficult to engage in goal-oriented behavior while experiencing anxiety.

Emotion regulation as predictor Novel theoretical frameworks emphasize that difficulties in emotion regulation are associated with the development and maintenance of anxiety disorders. Additionally, emotion regulation skills may be required to engage in and benefit from CBT. Furthermore, in an attempt to increase effectiveness, several newer treatments have included emotion regulation training in their treatments protocols.

The present study aims to examine attentional control and three facets of emotion regulation:

1. awareness and understanding of emotions,
2. acceptance of emotions, and
3. the ability to engage in goal-directed behavior, and refrain from impulsive behavior, when experiencing negative emotions as general predictors of outcome in CBT for anxiety disorders in a naturalistic, community-based mental health setting.

Our secondary aim is to examine a theoretical variables (i.e., socio-demographic data and clinical characteristics, such as comorbidity) as predictors of CBT outcome, as these have yet to be examined as predictors in real-world clinical settings in a mixed anxious sample.

Investigators expect that low ability to control attention will be associated with poorer treatment outcome. Similarly, it is expected that high scores on emotion dysregulation will be related to poorer treatment outcome. Given the exploratory nature of this study we will also be interested in testing non-linear relationships.

Method In order to maximize external validity, investigators are conducting the study within two real-world treatment clinics and employing minimal exclusion criteria recruiting a sample with mixed principal anxiety disorders. Patients will be recruited from the two clinics.

ELIGIBILITY:
Inclusion:

1. meet the diagnostic criteria for an anxiety disorder (social anxiety, generalized anxiety, panic disorder and agoraphobia) as primary diagnosis whether first episode or recurrent
2. are between 18 to 60 years of age
3. provide written informed consent
4. speak and understand Danish.

Exclusion:

1. cognitive disabilities (assessed with sub scales from Wechsler Adult Intelligence Scale Fourth-Edition, < 70)
2. alcohol or substance abuse (assessed during the preliminary consultations)
3. receiving any other psychotherapy during the study. Patients receiving medical treatment (e.g., antidepressants, Benzodiazepines) will also be included in the study and the treatment will be monitored closely.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with anxiety disorders from outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Beck Anxiety Inventory | 9 months
  Self-report questionnaire to assess level of anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Sara KK Nielsen, MSc, Principal Investigator — Department of Psychology
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Nielsen SK, Vangkilde S, Wolitzky-Taylor KB, Daniel SI, Hageman I. An investigation of general predictors for cognitive-behavioural therapy outcome for anxiety disorders in a routine clinical setting. BMJ Open. 2016 Mar 25;6(3):e010898. doi: 10.1136/bmjopen-2015-010898. PMID 27016248